CLINICAL TRIAL: NCT04071743
Title: A Randomized, Single-Center, Double-Blind, Parallel, Sham-Controlled Study of Gammacore Sapphire (Non-Invasive Vagus Nerve Stimulator) for the Acute and Preventive Treatment of Post-Traumatic Headache (GAP-PTH)
Brief Title: Study of Gammacore Sapphire for the Acute and Preventive Treatment of Post-Traumatic Headache (GAP-PTH)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary Investigator left UT Southwestern and was not replaced.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2019-0933
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Active Comparator): Treatment and Prevention with active gammacore device(vagus nerve stimulator)
  Interventions: Device: gammaCore Sapphire
- Sham (Sham Comparator): Treatment and Prevention with sham gammacore device(vagus nerve stimulator)
  Interventions: Device: sham gammaCore Sapphire

INTERVENTIONS:
Device: gammaCore Sapphire — non-invasive vagus nerve stimulator
  Arms: Treatment
Device: sham gammaCore Sapphire — sham gammaCore Sapphire
  Arms: Sham

SUMMARY:
The purpose of this single-center, prospective, randomized, double-blind, sham controlled, parallel-group study is to collect clinical data related to the safety and efficacy of vagus nerve stimulation for the acute and preventive treatment of Post Traumatic Headache.

DETAILED DESCRIPTION:
The study will enroll 60 subjects over a period of 14 weeks each. Subjects will use either a sham or active device to treat acute Post Traumatic Headache. Investigators will collect clinical data related to the use of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the ICHD-3 criteria for acute headache attributed to mild traumatic injury to the head
2. Experiences a minimum of 2 headaches (migraine or probable migraine phenotype) per week
3. Presentation to clinic between 2 and 4 weeks after injury
4. Able to provide written informed consent

Exclusion Criteria:

1. Any pre-existing primary headache disorder (with the exception of infrequent episodic tension type headache)
2. Any contraindication to using nVNS
3. Initiation or change in the dosage of any medication commonly used or headache prophylaxis 3 months before enrollment into the study
4. Continuous headache at the time of enrollment
5. PTH >4 weeks after injury
6. Structural abnormality at the nVNS treatment site (e.g., lymphadenopathy, previous surgery, abnormal anatomy)
7. Pain at the nVNS treatment site (e.g., dysesthesia, neuralgia, cervicalgia)
8. Other significant pain problem (e.g., cancer pain, fibromyalgia, other head or facial pain disorder) that, in the opinion of the Investigator, may confound the study assessments
9. Known or suspected severe cardiac disease (e.g., symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure) or an abnormal baseline electrocardiogram (ECG) within the last year (e.g., second- or third-degree heart block, prolonged QT interval, atrial fibrillation, atrial flutter, history of ventricular tachycardia or ventricular fibrillation, clinically significant premature ventricular contraction)
10. Known or suspected cerebrovascular disease (e.g., prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery)
11. Previous cervical vagotomy
12. A relative of or an employee of the Investigator or the clinical study site
13. Previously used gammaCore

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Relief of Post Traumatic Headache | Over 14 weeks
  Decrease in pain between active and sham treatment groups between the baseline assessment and 60 minutes post-treatment on a subset of questions from the Sport Concussion Assessment Tool, 5th edition (SCAT5) Graded Symptom Checklist

SECONDARY OUTCOMES:
Decrease in Pain | Over 14 weeks
  • Decrease in pain (based on the 7-point NRS) at 30 and 120 minutes after initial treatment, for all treated attacks in the nVNS and sham treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data outside of study

REFERENCES:
- [Background] Defrin R. Chronic post-traumatic headache: clinical findings and possible mechanisms. J Man Manip Ther. 2014 Feb;22(1):36-44. doi: 10.1179/2042618613Y.0000000053. PMID 24976746
- [Background] DiTommaso C, Hoffman JM, Lucas S, Dikmen S, Temkin N, Bell KR. Medication usage patterns for headache treatment after mild traumatic brain injury. Headache. 2014 Mar;54(3):511-9. doi: 10.1111/head.12254. PMID 24741687
- [Background] Lucas S. Posttraumatic Headache: Clinical Characterization and Management. Curr Pain Headache Rep. 2015 Oct;19(10):48. doi: 10.1007/s11916-015-0520-1. PMID 26280569
- [Background] Bree D, Levy D. Development of CGRP-dependent pain and headache related behaviours in a rat model of concussion: Implications for mechanisms of post-traumatic headache. Cephalalgia. 2018 Feb;38(2):246-258. doi: 10.1177/0333102416681571. Epub 2016 Dec 7. PMID 27899434
- [Background] Conidi FX. Interventional Treatment for Post-traumatic Headache. Curr Pain Headache Rep. 2016 Jun;20(6):40. doi: 10.1007/s11916-016-0570-z. PMID 27130542
- [Background] Packard RC. Treatment of chronic daily posttraumatic headache with divalproex sodium. Headache. 2000 Oct;40(9):736-9. doi: 10.1046/j.1526-4610.2000.00128.x. PMID 11091292
- [Background] Langdon R, Taraman S. Posttraumatic Headache. Pediatr Ann. 2018 Feb 1;47(2):e61-e68. doi: 10.3928/19382359-20180131-01. PMID 29446796
- [Background] Elahi F, Reddy C. High cervical epidural neurostimulation for post-traumatic headache management. Pain Physician. 2014 Jul-Aug;17(4):E537-41. PMID 25054404
- [Background] Schwedt TJ, Dodick DW, Hentz J, Trentman TL, Zimmerman RS. Occipital nerve stimulation for chronic headache--long-term safety and efficacy. Cephalalgia. 2007 Feb;27(2):153-7. doi: 10.1111/j.1468-2982.2007.01272.x. PMID 17257236
- [Background] Elahi F, Reddy C. Neuromodulation of the great auricular nerve for persistent post-traumatic headache. Pain Physician. 2014 Jul-Aug;17(4):E531-6. PMID 25054403
- [Background] Leung A, Fallah A, Shukla S, Lin L, Tsia A, Song D, Polston G, Lee R. rTMS in Alleviating Mild TBI Related Headaches--A Case Series. Pain Physician. 2016 Feb;19(2):E347-54. PMID 26815263
- [Background] Leung A, Metzger-Smith V, He Y, Cordero J, Ehlert B, Song D, Lin L, Shahrokh G, Tsai A, Vaninetti M, Rutledge T, Polston G, Sheu R, Lee R. Left Dorsolateral Prefrontal Cortex rTMS in Alleviating MTBI Related Headaches and Depressive Symptoms. Neuromodulation. 2018 Jun;21(4):390-401. doi: 10.1111/ner.12615. Epub 2017 May 30. PMID 28557049
- [Background] Howland RH. Vagus Nerve Stimulation. Curr Behav Neurosci Rep. 2014 Jun;1(2):64-73. doi: 10.1007/s40473-014-0010-5. PMID 24834378
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part I. Headache. 2016 Jan;56(1):71-8. doi: 10.1111/head.12647. Epub 2015 Sep 14. PMID 26364692
- [Background] Schachter SC. Vagus nerve stimulation therapy summary: five years after FDA approval. Neurology. 2002 Sep 24;59(6 Suppl 4):S15-20. doi: 10.1212/wnl.59.6_suppl_4.s15. PMID 12270963
- [Background] Cecchini AP, Mea E, Tullo V, Curone M, Franzini A, Broggi G, Savino M, Bussone G, Leone M. Vagus nerve stimulation in drug-resistant daily chronic migraine with depression: preliminary data. Neurol Sci. 2009 May;30 Suppl 1:S101-4. doi: 10.1007/s10072-009-0073-3. PMID 19415436
- [Background] Mauskop A. Vagus nerve stimulation relieves chronic refractory migraine and cluster headaches. Cephalalgia. 2005 Feb;25(2):82-6. doi: 10.1111/j.1468-2982.2005.00611.x. PMID 15658944
- [Background] Follesa P, Biggio F, Gorini G, Caria S, Talani G, Dazzi L, Puligheddu M, Marrosu F, Biggio G. Vagus nerve stimulation increases norepinephrine concentration and the gene expression of BDNF and bFGF in the rat brain. Brain Res. 2007 Nov 7;1179:28-34. doi: 10.1016/j.brainres.2007.08.045. Epub 2007 Aug 25. PMID 17920573
- [Background] Korley FK, Diaz-Arrastia R, Wu AH, Yue JK, Manley GT, Sair HI, Van Eyk J, Everett AD; TRACK-TBI investigators; Okonkwo DO, Valadka AB, Gordon WA, Maas AI, Mukherjee P, Yuh EL, Lingsma HF, Puccio AM, Schnyer DM. Circulating Brain-Derived Neurotrophic Factor Has Diagnostic and Prognostic Value in Traumatic Brain Injury. J Neurotrauma. 2016 Jan 15;33(2):215-25. doi: 10.1089/neu.2015.3949. Epub 2015 Sep 18. PMID 26159676
- [Background] Wurzelmann M, Romeika J, Sun D. Therapeutic potential of brain-derived neurotrophic factor (BDNF) and a small molecular mimics of BDNF for traumatic brain injury. Neural Regen Res. 2017 Jan;12(1):7-12. doi: 10.4103/1673-5374.198964. PMID 28250730
- [Background] Acheson A, Conover JC, Fandl JP, DeChiara TM, Russell M, Thadani A, Squinto SP, Yancopoulos GD, Lindsay RM. A BDNF autocrine loop in adult sensory neurons prevents cell death. Nature. 1995 Mar 30;374(6521):450-3. doi: 10.1038/374450a0. PMID 7700353
- [Background] Huang EJ, Reichardt LF. Neurotrophins: roles in neuronal development and function. Annu Rev Neurosci. 2001;24:677-736. doi: 10.1146/annurev.neuro.24.1.677. PMID 11520916
- [Background] Neren D, Johnson MD, Legon W, Bachour SP, Ling G, Divani AA. Vagus Nerve Stimulation and Other Neuromodulation Methods for Treatment of Traumatic Brain Injury. Neurocrit Care. 2016 Apr;24(2):308-19. doi: 10.1007/s12028-015-0203-0. PMID 26399249
- [Background] Lamb DG, Porges EC, Lewis GF, Williamson JB. Non-invasive Vagal Nerve Stimulation Effects on Hyperarousal and Autonomic State in Patients with Posttraumatic Stress Disorder and History of Mild Traumatic Brain Injury: Preliminary Evidence. Front Med (Lausanne). 2017 Jul 31;4:124. doi: 10.3389/fmed.2017.00124. eCollection 2017. PMID 28824913
- [Background] Silberstein SD, Calhoun AH, Lipton RB, Grosberg BM, Cady RK, Dorlas S, Simmons KA, Mullin C, Liebler EJ, Goadsby PJ, Saper JR; EVENT Study Group. Chronic migraine headache prevention with noninvasive vagus nerve stimulation: The EVENT study. Neurology. 2016 Aug 2;87(5):529-38. doi: 10.1212/WNL.0000000000002918. Epub 2016 Jul 13. PMID 27412146
- [Background] Tassorelli C, Grazzi L, de Tommaso M, Pierangeli G, Martelletti P, Rainero I, Dorlas S, Geppetti P, Ambrosini A, Sarchielli P, Liebler E, Barbanti P; PRESTO Study Group. Noninvasive vagus nerve stimulation as acute therapy for migraine: The randomized PRESTO study. Neurology. 2018 Jul 24;91(4):e364-e373. doi: 10.1212/WNL.0000000000005857. Epub 2018 Jun 15. PMID 29907608